CLINICAL TRIAL: NCT05061511
Title: Expression of Inflammasomes in Peri-implantitis and Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Principal Investigator, Prof Elena Calciolari, Ricercatore tipo B, University of Parma
Other Study IDs: P-003
Record Dates: First submitted 2021-05-27; First posted 2021-09-29 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis; Peri-Implantitis; Inflammation
MeSH Terms: conditions — Periodontitis; Peri-Implantitis; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gingival tissue will be collected in all 3 groups during surgical procedures such as periodontal surgeries, peri-implant surgeries, gingivectomies that the patients would undergo anyway, independently from taking part in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy gingival tissue: healthy patients with absence of gingivitis (full-mouth bleeding score <10%), no history of periodontal disease, having ≥20 teeth, and ≤1 tooth with interdental clinical attachment loss.
  Interventions: Other: Analysis of inflammasome expression; Other: Histological analysis
- Periodontitis patients: patients with stage III or IV periodontitis, which means that these patients would have deep periodontal lesions that extend at least to the mid portion of the roots and whose management is complicated by the presence of intrabony defects, furcation involvement, history of periodontal tooth loss and localized ridge defects.
  Interventions: Other: Analysis of inflammasome expression; Other: Histological analysis
- Peri-implantitis patients: patients affected by peri-implantitis, defined as radiographic evidence of bone loss ≥3 mm and probing pocket depth ≥6 mm around implants in conjunction with bleeding on probing; or defined as bleeding and/or suppuration on probing, increased probing pocket depth from a previous examination and loss of peri-implant bone.
  Interventions: Other: Analysis of inflammasome expression; Other: Histological analysis

INTERVENTIONS:
Other: Analysis of inflammasome expression — RNA isolation, spectrophotometric quantification, reverse transcription to cDNA and relative quantification of gene expression using a quantitative reverse transcription polymerase chain reaction (qRT-PCR). Specific inflammasome-related transcripts will be investigated, including ASC, caspase-1, IL-1beta, IL-18, NLRP3, NLRP2, AIM2, POP1, POP2, CARD16, CARD18, TRIM16, and TRIM20. A qRT-PCR System (e.g. StepOne Plus, Applied Biosystems) will be used for the amplification and analysis of the PCR products. Expression data will be reported as the ratio between each investigated target gene and GAPDH (used as housekeeping endogenous control).
Other: Histological analysis — gingival tissue samples will be prepared for paraffin inclusion and different stains will be used to evaluate the histological features of the tissues, distribution of inflammatory cells and alignment of collagen fibers.
  Moreover, a trained examiner will assess semi-quantitatively the inflammatory infiltrate under light microscopy.
  The expression of inflammatory/immune-related proteins such as NLRP3, ASC-2, IL-1beta and IL-18 protein expressions will be compared among the three groups by immunodetection methods

SUMMARY:
This is a laboratory-based study and it aims to evaluate the expression of inflammasomes in healthy gingiva and in the presence of peri-implantitis and periodontitis

DETAILED DESCRIPTION:
This is a laboratory-based study involving 48 systemically healthy patients divided into: healthy (H) (n=16), periodontitis stage III-IV (n=16) (PE) and peri-implantitis (n=16) (PI).

Patients will be recruited at the Centro di Odontoiatria, Dipartimento di Medicina e Chirurgia, Università di Parma.

Only 1 study visit will be performed, which coincides with the day in which the patient will receive the dental/gingival surgery.

After signing an informed consent form, all participants will undergo a full-mouth periodontal and peri-implant examination, including plaque index (FMPS), probing pocket depth (PPD), clinical attachment level (CAL), bleeding on probing (FMBS) recorded by a calibrated examiner from six sites per tooth/implant (mesiobuccal, midbuccal, distobuccal, distolingual, midlingual and mesiolingual) excluding third molars and using a manual University of North Carolina (UNC-15) periodontal probe. This is a routine examination done as part of dental assessments that allows to place a diagnosis of health, periodontitis or peri-implantitis.

Gingival tissue samples will be collected during surgical procedures such as gingivectomy, crown lengthening and resective surgery. In order to minimise the influence of bacteria from dental plaque as a source of local inflammation and preferentially evaluate the influence of systemic inflammatory conditions on the periodontal tissues, and following the standard of practice in periodontal and peri-implant treatment, patients belonging to the PE and PI group would have received non-surgical therapy and practical and theoretical sessions on general oral hygiene within 3 months before collecting the biopsy (Sanz et al., 2020).

Samples of the H group will be obtained from sites with gingival index (GI) <1 (Loe, 1967), no clinical attachment loss and without bleeding on probing. For PE and PI groups, tissue samples will be selected from the areas involved in the surgical procedure presenting the greatest level of inflammation and with the deepest PPD.

Each patient will contribute to one gingival tissue sample only, which may include up to 3 neighboring teeth/implants.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old

Exclusion Criteria:

* <18 years old
* Medical history that includes uncontrolled diabetes or hepatic or renal failure, or other serious medical conditions or transmittable diseases e.g. serious cardiovascular disease or AIDS.
* History of rheumatic fever, heart murmur, mitral valve prolapse, artificial heart valve or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
* Antibiotic, anti-inflammatory or anticoagulant therapy during the 2 weeks preceding the baseline exam.
* History of alcohol or drug abuse.
* In treatment with medications causing gingival overgrowth
* Smoking ≥10 cigarettes a day
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The definition of the 3 groups will be based on the features described by the 2017 World Workshop on the classification of periodontal and peri-implant conditions (Berglundh et al., 2018, Papapanou et al., 2018).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
difference in expression of inflammasome-related transcripts ASC, caspase-1, IL-1beta, IL-18, NLRP3, NLRP2, AIM2, POP1, POP2, CARD16, CARD18, TRIM16, and TRIM20 between the 3 groups | at the time of tissue collection (cross-sectional)

SECONDARY OUTCOMES:
Qualitative histological description of gingival tissue in the 3 groups | at the time of tissue collection (cross-sectional)
Semi-quantitative assessment of inflammatory score within histology sections | at the time of tissue collection (cross-sectional)
Differences in the expression of inflammatory-immune related proteins, such as NLRP3, ASC-2, IL-1beta and IL-18 proteins, as assessed by immunodetection methods in the 3 groups | at the time of tissue collection (cross-sectional)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitario di Odontoiatria, Parma, Italy

IPD SHARING:
Plan to Share IPD: No
Centro di Odontoiatria is the sponsor for this study. We will be using patient information in order to undertake this study and will act as the data controller for this study. This means that we are responsible for looking after patient information and using it properly. We will keep identifiable information for 20 years after the study has finished.
  The only people within the Centro di Odontoiatria who will have access to information that identifies the patients will be people who need to contact them about the research study, and make sure that relevant information about the study is recorded for their care, and to oversee the quality of the study or audit the data collection process. The people who analyse the information will not be able to identify patients and will not be able to find out their name or contact details.